CLINICAL TRIAL: NCT04736316
Title: Early Community Client-Led ART Delivery (CCLAD) to Optimize HIV Care Engagement in Nakivale Refugee Settlement
Brief Title: Early Community Client-LED ART Delivery in Nakivale Refugee Settlement
Acronym: Early CCLAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kelli O'Laughlin, Assistant Professor, School of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00008718; K23MH108440 (NIH)
Record Dates: First submitted 2020-07-27; First posted 2021-02-03 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: HIV Seropositivity
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early CCLAD (Experimental): Early community client-led ART delivery groups
  Interventions: Behavioral: Early CCLAD

INTERVENTIONS:
Behavioral: Early CCLAD — Community-based client led antiretroviral therapy delivery groups.

SUMMARY:
To pilot early community client-led ART (anti-retroviral therapy) delivery (CCLAD) in Nakivale Refugee Settlement in Uganda and assess the feasibility and acceptability of this intervention in this setting.

DETAILED DESCRIPTION:
Adults accessing routine HIV testing in Nakivale Refugee Settlement will be invited to participate. The study population will include adult refugees and Ugandan nationals of all genders older than 18 years of age. Pregnant women will be invited but Maternal Health Clinic will determine if they participate. Those that test positive for HIV will be invited to participate in the Early Community Client-Led ART Delivery group intervention.

Individuals will be offered research participation which will include an intake survey, an HIV test, and the option to participate in early community client-led ART delivery (early CCLAD) groups if diagnosed with HIV. Those interested in participating will have a consent form read aloud to them by a Research Assistant before being tested for HIV. Consent forms will be available in 4 languages: Runyankore, Kinyarwanda, Kiswahili and English, and will be read by multi-lingual Research Assistants. These individuals will be told at the outset that they can alternatively access free HIV testing at the outpatient department clinic if they prefer to not participate in any aspect of the research. After consent but prior to HIV testing, the investigators will conduct a baseline survey. This will include collection of contact information, demographic information, physical assessment, migration patterns, HIV testing history, perceived stigma, screening for mental disorders, and assessment of social support. Like the consent process, the survey will be available in 4 languages: Runyankore, Kinyarwanda, Kiswahili or English, and will be read aloud to participants with responses entered directly into a passcode-protected electronic tablet.

The first meeting of each Early CCLAD group will include an HIV clinic clinician. The first meeting is the one time in the intervention where participants will be compensated for their transportation to the clinic or to the meeting site (20,000 USH will be provided for each participant who attends this meeting). The HIV clinician, who will have been trained in the Early CCLAD group intervention, will help individuals in the group to understand their roles and responsibilities. The group will work together to plan future meeting dates and locations. The participants will decide if they would like to support the person responsible for picking up the ART each month (e.g. money, transportation, childcare, food). The participants will specify which dates they will be responsible to attend HIV clinic and pick up ART for the group. They will discern if they would like to identify a connecting activity to be integrated into their group (e.g. exercise, faith, livelihood, craft). The participant group will select a Team Leader to coordinate communication between the group and the healthcare facility. Finally, an important part of this first meeting is that the HIV clinician will conduct a standard comprehensive clinical exam and will refer each person/participant for any necessary laboratory testing.

Monthly "Early CCLAD" meetings: The "Early CCLAD" intervention will require monthly group meetings. This is intentionally more frequent than is suggested in the Ugandan Ministry of Health guidelines (which recommends visits every 3 months) as this intervention will occur at the time of diagnosis rather than when a person is deemed "stable" in care. Before the designated individual goes to clinic in any given month, they will be responsible for connecting with each group member to ask about how they are feeling and to see if they have any questions to ask of the HIV clinic staff. That individual will then attend HIV clinic and communicate about the status of each group member. They will collect information from the clinic and pre-packed ART for each group member. The "Early CCLAD" group will then meet at their predetermined location so that the individual who attended clinic can share information from the clinic and can distribute the ART to each person in the group. If a participant misses a CCLAD group, they can present to the HIV clinic to pick up their ART refill if a member of the group cannot arrange delivery or pickup.

Additional clinic attendance: All participants assigned to an "Early CCLAD" group will be expected to attend HIV clinic in person twice yearly for a clinical evaluation and a viral load check. The HIV clinician will work with the team to decide if they prefer their twice annual HIV clinic visits on the same day but individually, on the same day as a group, or individually on different schedules from others in the group. Additionally, individuals will attend clinic in person when they do not feel well, when they have any questions they prefer to ask the clinicians directly, when additional laboratory testing is required, and when requested by HIV clinic staff to optimize their medical care. In cases where the participants are deemed clinically unstable and are in need of regular clinical follow up (e.g. develops an opportunistic infection, develops other co-morbidity, has a viral load > 1,000 copies/mL), clients will be asked to attend the clinic monthly with the rotating group member collecting group ART refill or to step in as the group member responsible for attending clinic that month. Individuals "Up referred" by HIV clinic staff to monthly HIV clinic visits should still participate in the "Early CCLAD" groups to receive psychosocial support and other benefits of community group care.

Option to stop the "Early CCLAD" group at any time: Participants can opt to stop Early CCLAD participation at any time. If willing, they will be asked to participate in a brief exit interview so the investigators can better understand what aspects of the intervention were acceptable or not acceptable to them.

"Early CCLAD" groups and HIV clinic connectedness: To ensure the Early CCLAD intervention participants remain well integrated into HIV clinic, the research staff will meet regularly with the HIV clinic staff to update them on the intervention and to discuss specific problems and specific individuals needing specialized care. Additionally, efforts will be made so that participant HIV clinic files and pre-packed medications are ready for the visit of the individual Early CCLAD group member each month. Finally, participants will be reminded frequently that they are expected and welcome to attend clinic when they do not feel well or when they have any questions or needs that are not being met through group care.

Follow-up data collection: Early CCLAD group participants will be given components of the intake survey (i.e. to assess mental health screening, perceived stigma, and social support) again 6-months after they began participation in the intervention. Some of this may occur in an interview setting which is recorded and then later transcribed. Additionally, data will be collected to assess retention in group care, ART medication pick-up, and HIV clinic outcomes.

ELIGIBILITY:
Inclusion Criteria:

• Adults ≥ 18 years of age who present to the Nakivale Health Center and agree/consent to test for HIV.

Exclusion Criteria:

* Unable to understand one of the study languages (English, Kinyarwanda, Kiswahili, Runyankore).
* Subjects who do not test positive for HIV at health center will not be eligible to participate in the early community-based client-led antiretroviral therapy delivery intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli N O'Laughlin, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Nakivale Refugee Settlement, Isingiro, Uganda

IPD SHARING:
Plan to Share IPD: No
Pilot research findings will be shared in a peer-reviewed journal. Additional research data sharing requests will be considered by the PI.

RESULTS

PARTICIPANT FLOW:
Groups:
- Early CCLAD Participants: Subjects receiving Early CCLAD intervention
- Non Early CCLAD Participants: As this was the pilot study/feasibility trial, the study design was not intended to compare the intervention group to a control group. This pilot study did not have a control group. This group represents subjects not receiving the Early CCLAD intervention. Although they were initially eligible, they were unable to be enrolled for a variety of reasons, such as distance to clinic or not living close to other Early CCLAD group members. We provide this data to compare pilot study participants to non-participants, not as a control group.
Period: Overall Study
Arm/Group | Early CCLAD Participants | Non Early CCLAD Participants
Started | 31 | 61
Completed | 31 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Early CCLAD Participants: Subjects receiving CCLAD intervention
- Non Early CCLAD Participants: As this was the pilot study/feasibility trial, the study design was not intended to compare the intervention group to a control group. This pilot study did not have a control group. This group represents subjects not receiving the Early CCLAD intervention. Although they were initially eligible, they were unable to be enrolled for a variety of reasons, such as distance to clinic or not living close to other Early CCLAD group members. We provide this demographic data to compare pilot study participants to non-participants, not as a control group.
- Total: Total of all reporting groups
Arm/Group | Early CCLAD Participants | Non Early CCLAD Participants | Total
Number analyzed (Participants) | 31 | 61 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (10.4) | 31.9 (10.3) | 33.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 38 | 53
  Male | 16 | 23 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 61 | 92
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Refugees [Count of Participants; unit: Participants] | 21 | 19 | 40
Education [Count of Participants; unit: Participants]
  No School | 7 | 11 | 18
  Some Primary School | 17 | 30 | 47
  Completed Primary School | 2 | 9 | 11
  Beyond Primary School | 5 | 11 | 16
Willingness to particpate in an Early CCLAD group, n(%) [Count of Participants; unit: Participants] | 31 | 43 | 74
Mental Health Conditions [Count of Participants; unit: Participants]
  Anxiety | 15 | 19 | 34
  Depression | 15 | 22 | 37
  Low Social Support | 5 | 4 | 9
  PTSD | 20 | 38 | 58
Self-Reported Health Status [Count of Participants; unit: Participants] — Participants self-reported their health status by responding to the prompt: "In general, would you say your health is excellent, very good, good, fair or poor?" Subjects chose one of seven answer options provided: "Excellent, very good, good, fair, poor, do not know, no answer"
  Participants
    Fair/Poor | 16 | 33 | 49
    Good/Very Good | 15 | 28 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in HIV Care (Linkage) Among the Early CCLAD Participants
Description: Attendance in one Early CCLAD group meeting (yes/no)
Time Frame: Within 90 days of study initiation excluding the day of diagnosis
Population: Data was not collected from the "Non Early CCLAD Participants"
Measure: Count of Participants; unit: Participants
Arm/Group | Early CCLAD Participants
Number analyzed (Participants) | 31
Participants | 31

2. Primary Outcome: Number of Early CCLAD Group Visits Attended (Retention) Among Early CCLAD Participants
Description: Attendance in monthly Early CCLAD group meetings (yes/no). With an intention to treat, description of how many monthly group meetings were attended in the first 6 months of the intervention including Early CCLAD community visits, but not including HIV clinic visits
Time Frame: 6 months
Population: Data was not collected from the "Non Early CCLAD Participants"
Measure: Mean (Inter-Quartile Range); unit: Early CCLAD group visits
Arm/Group | Early CCLAD Participants
Number analyzed (Participants) | 31
Early CCLAD group visits | 3.3 [2 to 5]

3. Primary Outcome: ART Initiation
Description: Number of participants who picked up anti-retroviral therapy (ART) at least once over the 6 month period as documented in the written HIV clinic record
Time Frame: 6 months
Population: As this was the pilot study/feasibility trial, the study design was not intended to compare the intervention group to a control group. This pilot study did not have a control group. Data was not collected from the "Non Early CCLAD Participants"
Measure: Count of Participants; unit: Participants
Arm/Group | Early CCLAD Participants
Number analyzed (Participants) | 31
Participants | 31

4. Primary Outcome: Clinical Outcomes: Number of Participants With Viral Suppression
Description: Viral suppression defined by <1000 copies/mL or CD4 count >250 cells/mm3 as documented in the HIV clinic records
Time Frame: 6 month period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Early CCLAD Participants
Number analyzed (Participants) | 31
Participants
  Virally Suppressed (VL <1000 or CD4>250) | 20
  Not Virally Suppressed (VL≥1000 or CD4≤250) | 3
  Missing Clinical Data | 8

5. Primary Outcome: Total Number of Clinic Visits Per Participant (Incl. CCLAD Visits)
Description: All clinic and CCLAD visits per participant
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Inter-Quartile Range); unit: visits
Arm/Group | Early CCLAD Participants
Number analyzed (Participants) | 31
visits | 5.1 [4 to 6]

6. Primary Outcome: Survey Score Related to Psychosocial Factors: Perceived Health
Description: Question: "In general, would you say your health is excellent, very good, good, fair or poor?" Answer options: "Excellent, very good, good, fair, poor, do not know, no answer" This is among participants who completed both baseline and follow-up surveys only.
Time Frame: baseline survey and 6 month follow-up survey
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Early CCLAD Participants
Number analyzed (Participants) | 21
Participants
  Baseline: Fair/Poor | 11
  Baseline: Good/Very Good | 10
  6 Month Follow-Up: Fair/Poor | 5
  6 Month Follow-Up: Good/Very Good | 16

7. Primary Outcome: Survey Score Related Factors: Screened Positive for Depression
Description: Depression measured via Patient health questionnaire depression assessment (PHQ-9); 9 questions with 0-3 score for each answer. Interpretation of score: 0-4= minimal or no depression; 5-9= mild depression; 10-14=moderate depression. For this study, we considered a positive screen for depression as a PHQ-9 score of >=10.
  This analysis includes only those who participated in baseline and 6 month surveys.
Time Frame: baseline and 6 month surveys
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Early CCLAD Participants
Number analyzed (Participants) | 21
Participants
  Baseline | 10
  6 Month Follow-Up | 4

8. Primary Outcome: Survey Score Related Factors: Screened Positive for Anxiety
Description: Anxiety measured via Generalized anxiety disorder (GAD-7) tool; 7 questions with 0-3 score for each answer; Interpretation of total score: 0-4=minimal anxiety; 5-9= mild anxiety; 10-14=moderate anxiety; 15-21=severe anxiety. For this study, those with a score of >= 10 were considered to have screened in for anxiety.
  This analysis includes only those who participated in baseline and 6 month surveys.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Early CCLAD Participants
Number analyzed (Participants) | 21
Participants
  Baseline | 9
  6 Month Follow-Up | 6

9. Primary Outcome: Survey Score Related Factors: Screening Positive for PTSD
Description: PTSD measured via Post-traumatic stress disorder (PCL-6) scale; 6 questions with 1-5 score for each question; Interpretation of Total score: greater than or equal to 14 is a positive screen.
  This analysis includes only those who participated in baseline and 6 month surveys.
Time Frame: baseline and 6 month surveys
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Early CCLAD Participants
Number analyzed (Participants) | 21
Participants
  Baseline | 12
  6 Month Follow-Up | 9

10. Primary Outcome: Survey Score Related Factors: Screening Positive for Low of Social Support
Description: Social Support measured via Social support (BS6) scale; 6 questions with scores 1-4 for each answer; Interpretation of total score: 6-11= low (a positive screen for lack of social support), 12-17=moderate (at least occasional support); 18-23= high; 24=very high (maximum, always supported). For this study we considered <= 11 as a positive screen for low of social support.
  This analysis includes only those who participated in baseline and 6 month surveys.
Time Frame: baseline and 6 month surveys
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Early CCLAD: Subjects receiving Early CCLAD intervention
Arm/Group | Early CCLAD
Number analyzed (Participants) | 21
Participants
  baseline | 4
  6 month survey | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participants from the date of enrollment until they finished study activities. This was a maximum period of 1 year and 9 months.
Arm/Group | Early CCLAD Participants | Non Early CCLAD Participants
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/61
Other Adverse Events (participants affected / at risk) | 0/31 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT04736316/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT04736316/SAP_001.pdf